CLINICAL TRIAL: NCT01722331
Title: A 64-Week, Phase 3, Randomized, Placebo-Controlled, Parallel Design Study to Evaluate the Efficacy and Safety/Tolerability of Subcutaneous Tildrakizumab (SCH 900222/MK-3222), Followed by an Optional Long-Term Safety Extension Study, in Subjects With Moderate-to-Severe Chronic Plaque Psoriasis (Protocol No. MK-3222-010)
Brief Title: A Study to Evaluate the Efficacy and Safety of Subcutaneous MK-3222, Followed by an Optional Long-Term Safety Extension Study, in Participants With Moderate-to-Severe Chronic Plaque Psoriasis (MK-3222-010)
Acronym: reSURFACE 1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3222-010; 2012-002255-42 (EudraCT Number); P07770 (Other: Merck Protocol Number); 132284 (Registry Identifier: JAPIC-CTI)
Record Dates: First submitted 2012-11-02; First posted 2012-11-06 (Estimated); Results first posted 2018-06-13 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — tildrakizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Tildrakizumab 200 mg (Experimental): Tildrakizumab 200 mg administered subcutaneously (SC) once a week at Weeks 0 and 4 and then every 12 weeks.
  Interventions: Drug: Tildrakizumab 200 mg; Drug: Matching Placebo
- Tildrakizumab 100 mg (Experimental): Tildrakizumab 100 mg administered SC once a week at Weeks 0 and 4 and then every 12 weeks.
  Interventions: Drug: Tildrakizumab 100 mg; Drug: Matching Placebo
- Placebo (Placebo Comparator): Matching placebo administered SC once a week at Weeks 0 and 4.
  Interventions: Drug: Tildrakizumab 200 mg; Drug: Tildrakizumab 100 mg; Drug: Matching Placebo

INTERVENTIONS:
Drug: Tildrakizumab 200 mg — Two tildrakizumab 100 mg/mL pre-filled syringes (PFS)
  Other Names: MK-3222, SCH 900222
  Arms: Placebo; Tildrakizumab 200 mg
Drug: Tildrakizumab 100 mg — Tildrakizumab 100 mg/mL PFS
  Other Names: MK-3222, SCH 900222
  Arms: Placebo; Tildrakizumab 100 mg
Drug: Matching Placebo — Matching placebo to tildrakizumab PFS

SUMMARY:
This study is being conducted to evaluate the efficacy and safety/tolerability of subcutaneous tildrakizumab (MK-3222), followed by an optional long-term safety extension study, in participants with moderate-to-severe chronic plaque psoriasis.

DETAILED DESCRIPTION:
Participants are initially randomized to receive tildrakizumab 200 or 100 mg once weekly at Weeks 0, 4, and every 12 weeks thereafter; or placebo at Weeks 0 and 4.

At Week 12, participants initially randomized to placebo will be re-randomized to receive either tildrakizumab 200 or 100 mg at Weeks 12 and 16.

At Week 28, all participants enrolled will be assessed for their improvement in PASI score from baseline.

RESPONDERS: Participants initially randomized to tildrakizumab who achieve at least a 75% improvement from baseline PASI will be re-randomized to either continue on their initial treatment or to receive placebo at Week 28.

* Participants who are re-randomized to continue on their initial treatment will continue tildrakizumab 200 or 100 mg every 12 weeks through Week 64.
* Participants who are re-randomized to placebo will receive placebo every 4 weeks until relapse (reduction in maximum PASI response by 50%). If relapse occurs, the tildrakizumab dose that the participants was originally randomized to at baseline will be re-initiated (tildrakizumab 200 or 100 mg). Participants will be dosed tildrakizumab at the visit when the relapse occurs, and subsequent dosing of tildrakizumab will be given 4 weeks after treatment re-initiation, and every 12 weeks thereafter through Week 64.

PARTIAL RESPONDERS: Participants initially randomized to tildrakizumab who achieved a PASI response of ≥50% but <75% improvement from baseline will be assigned a treatment regimen as described below, with their first dose started at Week 28.

* Participants initially randomized to tildrakizumab 200 mg will remain on tildrakizumab 200 mg every 12 weeks.
* Participants initially randomized to tildrakizumab 100 mg will be re-randomized to either remain on tildrakizumab 100 mg every 12 weeks or to receive tildrakizumab 200 mg every 12 weeks.
* Participants initially randomized to placebo who achieved ≥50% improvement from baseline in PASI will receive tildrakizumab (200 or 100 mg) according to their re-randomized treatment assignment at Week 12 and continue on this treatment every 12 weeks through Week 64.

NON-RESPONDERS: Participants who did not achieve at least 50% improvement from baseline PASI at Week 28 will be discontinued from the study.

EXTENSION: Participants will receive tildrakizumab 200 mg or 100 mg every 12 weeks through Extension Week 192, depending on the treatment received at the time of completion of the base study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of moderate-to-severe plaque psoriasis for at least 6 months prior to study enrollment
* A candidate for phototherapy or systemic therapy
* For the extension study: must have completed Part 3 of the base study
* For the extension study: must have achieved at least a PASI-50 response by the end of Part 3 of the base study
* For the extension study: must have received active tildrakizumab (MK-3222) treatment within 12 weeks prior to the end of Part 3 of the base study
* Premenopausal female participants must agree to abstain from heterosexual activity or use a medically accepted method of contraception or use appropriate effective contraception as per local regulations or guidelines
* If enrolled at a Japanese site, participants with psoriatic arthritis using non-steroidal anti-inflammatory drugs (NSAIDs) must be on a stable dose for at least 4 weeks prior to the first dose of study drug and must not be expected to require an increase in dose over the course of the study

Exclusion Criteria:

* Has erythrodermic psoriasis, predominantly pustular psoriasis, medication-induced or medication-exacerbated psoriasis, or new onset guttate psoriasis
* Current or history of severe psoriatic arthritis and is well-controlled on current treatment
* Women of child-bearing potential who are pregnant, intend to become pregnant within 6 months of completing the trial, or who are breast feeding
* Expected to require topical treatment, phototherapy, or systemic treatment during the trial
* Presence of any infection
* History of recurrent infection requiring treatment with systemic antibiotics within 2 weeks of screening
* Previous use of tildrakizumab (MK-3222) or other IL-23/Th-17 pathway inhibitors including P40, p19, and IL-17 antagonists
* Evidence of active or untreated latent tuberculosis (TB)
* Positive test for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV)
* At Japanese sites, positive test for HBs antibody and hepatitis B virus (HBV) deoxyribonucleic acid (DNA)
* At Japanese sites, positive test for the Hepatitis B core (HBc) antibody and HBV DNA
* For the extension study: women of child-bearing potential who are pregnant, intend to become pregnant within 6 months of completing the trial, or who are breast feeding
* For the extension study: active or uncontrolled significant organ dysfunction or clinically significant laboratory abnormalities
* For the extension study: expected to require topical treatment, phototherapy, or systemic treatment during the extension study
* At Japanese sites, abnormal for Beta D Glucan and/or KL-6 test result(s) at the screening visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 772 (Actual)
Dates: Start 2012-12-06 (Actual); Primary Completion 2015-10-28 (Actual); Study Completion 2021-11-10 (Actual)

REFERENCES:
- [Result] Reich K, Papp KA, Blauvelt A, Tyring SK, Sinclair R, Thaci D, Nograles K, Mehta A, Cichanowitz N, Li Q, Liu K, La Rosa C, Green S, Kimball AB. Tildrakizumab versus placebo or etanercept for chronic plaque psoriasis (reSURFACE 1 and reSURFACE 2): results from two randomised controlled, phase 3 trials. Lancet. 2017 Jul 15;390(10091):276-288. doi: 10.1016/S0140-6736(17)31279-5. Epub 2017 Jun 6. PMID 28596043
- [Derived] Armstrong AW, Blauvelt A, Lebwohl M, Asahina A, Gogineni R, Griffiths CEM. Efficacy and safety of tildrakizumab in patients with early- vs. late-onset psoriasis. Br J Dermatol. 2025 Aug 18;193(3):442-450. doi: 10.1093/bjd/ljaf171. PMID 40365708
- [Derived] Thaci D, Gerdes S, Du Jardin KG, Perrot JL, Puig L. Efficacy of Tildrakizumab Across Different Body Weights in Moderate-to-Severe Psoriasis Over 5 Years: Pooled Analyses from the reSURFACE Pivotal Studies. Dermatol Ther (Heidelb). 2022 Oct;12(10):2325-2341. doi: 10.1007/s13555-022-00793-z. Epub 2022 Sep 13. PMID 36098877
- [Derived] Igarashi A, Nakagawa H, Morita A, Okubo Y, Sano S, Imafuku S, Tada Y, Honma M, Mendelsohn AM, Kawamura M, Ohtsuki M. Efficacy and safety of tildrakizumab in Japanese patients with moderate to severe plaque psoriasis: Results from a 64-week phase 3 study (reSURFACE 1). J Dermatol. 2021 Jun;48(6):853-863. doi: 10.1111/1346-8138.15789. Epub 2021 Feb 25. PMID 33630387
- [Derived] Kerbusch T, Li H, Wada R, Jauslin PM, Wenning L. Exposure-response characterisation of tildrakizumab in chronic plaque psoriasis: Pooled analysis of 3 randomised controlled trials. Br J Clin Pharmacol. 2020 Sep;86(9):1795-1806. doi: 10.1111/bcp.14280. Epub 2020 Mar 25. PMID 32162721
- [Derived] Elewski B, Menter A, Crowley J, Tyring S, Zhao Y, Lowry S, Rozzo S, Mendelsohn AM, Parno J, Gordon K. Sustained and continuously improved efficacy of tildrakizumab in patients with moderate-to-severe plaque psoriasis. J Dermatolog Treat. 2020 Dec;31(8):763-768. doi: 10.1080/09546634.2019.1640348. Epub 2019 Jul 22. PMID 31268369
- [Derived] Reich K, Warren RB, Iversen L, Puig L, Pau-Charles I, Igarashi A, Ohtsuki M, Falques M, Harmut M, Rozzo S, Lebwohl MG, Cantrell W, Blauvelt A, Thaci D. Long-term efficacy and safety of tildrakizumab for moderate-to-severe psoriasis: pooled analyses of two randomized phase III clinical trials (reSURFACE 1 and reSURFACE 2) through 148 weeks. Br J Dermatol. 2020 Mar;182(3):605-617. doi: 10.1111/bjd.18232. Epub 2019 Jul 18. PMID 31218661
- [Derived] Jauslin P, Kulkarni P, Li H, Vatakuti S, Hussain A, Wenning L, Kerbusch T. Population-Pharmacokinetic Modeling of Tildrakizumab (MK-3222), an Anti-Interleukin-23-p19 Monoclonal Antibody, in Healthy Volunteers and Subjects with Psoriasis. Clin Pharmacokinet. 2019 Aug;58(8):1059-1068. doi: 10.1007/s40262-019-00743-7. PMID 30915660

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The tables below present the Participant Flow for the Base Study only (Weeks 0 to 64: Part 1 for 12 weeks, Part 2 for 16 weeks, and Part 3 for 36 weeks).
Groups:
- Tildrakizumab 200 mg (Parts 1, 2 & 3): Tildrakizumab 200 mg administered subcutaneously (SC) once a week at Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28, 40, 52 and 64 (Part 3).
- Tildrakizumab 100 mg (Parts 1, 2 & 3): Tildrakizumab 100 mg administered SC once a week at Weeks 0 and 4 (Part 1), Week 16 (Part 2), and Weeks 28, 40, 52 and 64 (Part 3).
- Tildrakizumab 100 mg (Parts 1 & 2): Tildrakizumab 100 mg administered SC once a week at Weeks 0 and 4 (Part 1) and Week 16 (Part 2).
- Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3): Tildrakizumab 100 mg administered SC once a week at Weeks 0 and 4 (Part 1) and Week 16 (Part 2). Tildrakizumab 200 mg administered SC once a week at Weeks 28, 40, 52, and 64 (Part 3).
- Placebo (Part 1): Matching placebo administered SC once a week at Weeks 0 and 4 (Part 1).
- Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3): Matching placebo administered SC once a week at Weeks 0 and 4 (Part 1). Tildrakizumab 200 mg administered SC once a week at Week 16 (Part 2) and Weeks 28, 40, 52 and 64 (Part 3).
- Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3): Matching placebo administered SC once a week at Weeks 0 and 4. Tildrakizumab 200 mg administered SC once a week at Week 16 (Part 2) and Weeks 28, 40, 52 and 64 (Part 3).
Period: Part 1
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) | Tildrakizumab 100 mg (Parts 1, 2 & 3) | Tildrakizumab 100 mg (Parts 1 & 2) | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) | Placebo (Part 1) | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3)
Started | 308 | 249 | 41 | 19 | 9 | 72 | 74
Completed | 298 | 249 | 32 | 19 | 0 | 72 | 74
Not Completed | 10 | 0 | 9 | 0 | 9 | 0 | 0
Not completed — Adverse Event | 5 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 2 | 0 | 1 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 3 | 0 | 1 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Progressive Disease | 0 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 3 | 0 | 3 | 0 | 0
Period: Part 2
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) | Tildrakizumab 100 mg (Parts 1, 2 & 3) | Tildrakizumab 100 mg (Parts 1 & 2) | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) | Placebo (Part 1) | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3)
Started | 298 | 249 | 31 (1 participant who completed Part 1 did not enter Part 2) | 19 | 0 | 72 | 74
Completed | 279 | 249 | 0 | 19 | 0 | 62 | 67
Not Completed | 19 | 0 | 31 | 0 | 0 | 10 | 7
Not completed — Adverse Event | 3 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lack of Efficacy | 3 | 0 | 11 | 0 | 0 | 3 | 3
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0 | 1 | 1
Not completed — Non-Compliance with Study Drug | 1 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 2 | 0 | 0 | 0 | 0
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Progressive Disease | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 3 | 0 | 0 | 2 | 2
Not completed — Other Protocol Specified Criteria | 6 | 0 | 10 | 0 | 0 | 2 | 1
Period: Part 3
Arm/Group | Tildrakizumab 200 mg (Parts 1, 2 & 3) | Tildrakizumab 100 mg (Parts 1, 2 & 3) | Tildrakizumab 100 mg (Parts 1 & 2) | Tildrakizumab 100 mg (Parts 1 & 2)/ 200 mg (Part 3) | Placebo (Part 1) | Placebo (Part 1)/ Tildrakizumab 200 mg (Parts 2 & 3) | Placebo (Part 1)/ Tildrakizumab 100 mg (Parts 2 & 3)
Started | 279 | 249 | 0 | 19 | 0 | 62 | 67
Completed | 264 | 232 | 0 | 18 | 0 | 59 | 65
Not Completed | 15 | 17 | 0 | 1 | 0 | 3 | 2
Not completed — Adverse Event | 2 | 2 | 0 | 1 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 3 | 4 | 0 | 0 | 0 | 1 | 0
Not completed — Non-Compliance with Study Drug | 0 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 1 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 2 | 1 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 4 | 7 | 0 | 0 | 0 | 2 | 1
Not completed — Other Protocol Specified Criteria | 1 | 1 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Overall Number of Baseline Participants includes randomized participants according to assigned treatment for Part 1 of the study.
Groups:
- Tildrakizumab 200 mg (Part 1): Tildrakizumab 200 mg administered subcutaneously (SC) once a week at Weeks 0 and 4 and then every 12 weeks.
- Tildrakizumab 100 mg (Part 1): Tildrakizumab 100 mg administered SC once a week at Weeks 0 and 4 and then every 12 weeks.
- Placebo (Part 1): Matching placebo administered SC once a week at Weeks 0 and 4.
- Total: Total of all reporting groups
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1) | Total
Number analyzed (Participants) | 308 | 309 | 155 | 772
Age, Continuous [Mean (Standard Deviation); unit: Years] | 46.9 (13.16) | 46.4 (13.09) | 47.9 (13.55) | 46.9 (13.21)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 102 | 55 | 239
  Male | 226 | 207 | 100 | 533
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 37 | 34 | 19 | 90
  Not Hispanic or Latino | 271 | 275 | 135 | 681
  Unknown or Not Reported | 0 | 0 | 1 | 1
Physician's Global Assessment (PGA) score [Count of Participants; unit: Participants] — The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration; 1= Minimal; 2 =Mild; 3= Moderate; 4= Marked; 5= Severe. Round average to the nearest whole number. Population: Analysis population includes participants with baseline PGA data.
  Participants
    number analyzed (Participants) | 308 | 309 | 154 | 771
    <3 | 0 | 1 | 0 | 1
    3 | 202 | 206 | 111 | 519
    4 | 95 | 95 | 41 | 231
    5 | 11 | 7 | 2 | 20
Body weight [Count of Participants; unit: Participants]
  <=90 kg | 182 | 183 | 93 | 458
  >90 kg | 126 | 126 | 62 | 314
Prior exposure to biologics therapy for psoriasis [Count of Participants; unit: Participants] — The following therapies constitute biologics therapy for psoriasis: efalizumab, alefacept, infliximab, adalimumab, ustekinumab, and etanercept.
  Participants
    Yes | 71 | 71 | 35 | 177
    No | 237 | 238 | 120 | 595

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Psoriasis Area Sensitivity Index 75 (PASI-75) Response at Week 12 (Base Study)
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the amount of body surface for each region involved (head=0.1; upper limbs=0.2; trunk= 0.3; and lower limbs=0.4) and the degree of involvement for each body region (0=no involvement to 6=90-100% involvement). Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-75 response indicates the number of participants achieving a 75% reduction in PASI score compared to baseline.
Time Frame: Week 12 (or end of trial if prior to Week 12)
Population: Analysis population consists of all randomized participants who received at least one dose of assigned study drug between Weeks 0 and 12.
Measure: Number; unit: Percentage of Participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Percentage of Participants | 62.3 | 63.8 | 5.8
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; Stratified by body weight (<=90kg, >90kg) and prior exposure to biologic therapy for psoriasis (yes/no). P-values are not adjusted for multiplicity; Difference in percentages = 56.6, 95% CI 2-sided [49.6 to 62.8]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 58.0, 95% CI 2-sided [51.0 to 64.1]

2. Primary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) Score of Clear or Minimal With at Least a 2 Grade Reduction From Baseline at Week 12 (Base Study)
Description: The PGA is used to determine the overall severity of a participant's psoriasis lesions at a given time point. Overall lesions will be graded for thickness, erythema, and scaling on a scale from 0 to 5. The sum of the 3 scales will be divided by 3 to obtain the PGA score. PGA is assessed as: 0= Cleared, except for residual discoloration. 1= Minimal, majority of lesions have individual scores that average 1. 2 =Mild, majority of lesions have individual scores that average 2. 3= Moderate, majority of lesions have individual scores that average 3. 4= Marked, majority of lesions have individual scores that average 4. 5= Severe, majority of lesions have individual scores that average 5.
Time Frame: Baseline and Week 12 (or end of trial if prior to Week 12)
Population: as for outcome 1
Measure: Number; unit: Percentage of Participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Percentage of Participants | 59.1 | 57.9 | 7.1
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 52.1, 95% CI 2-sided [44.8 to 58.5]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 50.9, 95% CI 2-sided [43.6 to 57.4]

3. Primary Outcome: Number of Participants Experiencing an Adverse Event Up to Week 12 (Base Study)
Description: An adverse event is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment.
Time Frame: Up to 12 weeks
Population: Analysis population included all randomized participants who received at least 1 dose of study medication during Weeks 0 to 12 based on the treatment actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Participants | 130 | 146 | 74

4. Primary Outcome: Number of Participants Discontinuing Study Drug Due to an Adverse Event Up to Week 12 (Base Study)
Description: as for outcome 3
Time Frame: Up to 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Participants | 5 | 0 | 1

5. Primary Outcome: Number of Participants Discontinuing Study Drug Due to a Drug-Related Adverse Event (Base Study)
Description: A drug-related adverse event is an adverse event that has been determined by the investigator to be related to the study drug.
Time Frame: Up to 12 weeks
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Participants | 2 | 0 | 0

6. Secondary Outcome: Percentage of Participants With PASI-90 Response At Week 12
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the amount of body surface for each region involved (head=0.1; upper limbs=0.2; trunk= 0.3; and lower limbs=0.4) and the degree of involvement for each body region (0=no involvement to 6=90-100% involvement). Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-90 response indicates the number of participants achieving a 90% reduction in PASI score compared to baseline.
Time Frame: Week 12 (or end of trial if prior to Week 12)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Percentage of participants | 35.4 | 34.6 | 2.6
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 32.9, 95% CI 2-sided [26.8 to 38.8]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 32.1, 95% CI 2-sided [25.9 to 38.0]

7. Secondary Outcome: Percentage of Participants With PASI-100 Response at Week 12
Description: The PASI is a measure of the average redness, thickness, and scaliness of lesions (each graded on a 0-4 scale), weighed by the amount of body surface for each region involved (head=0.1; upper limbs=0.2; trunk= 0.3; and lower limbs=0.4) and the degree of involvement for each body region (0=no involvement to 6=90-100% involvement). Calculated PASI score ranges from 0 to 72, with higher score indicating more severe disease status. The PASI-100 response indicates the number of participants achieving a 100% reduction in PASI score compared to baseline.
Time Frame: Week 12 (or end of trial if prior to Week 12)
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Percentage of participants | 14.0 | 13.9 | 1.3
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 12.7, 95% CI 2-sided [8.3 to 17.2]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg (Part 1) vs Placebo (Part 1); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 12.7, 95% CI 2-sided [8.0 to 17.3]

8. Secondary Outcome: Baseline Dermatology Life Quality Index (DLQI) Score
Description: The DLQI questionnaire consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life.
Time Frame: Baseline
Population: Analysis population consists of all randomized participants who received at least one dose of assigned study drug between Weeks 0 and 12 and have baseline DLQI measurement
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Score on a scale | 13.2 (6.87) | 13.9 (6.68) | 13.2 (7.25)

9. Secondary Outcome: Change From Baseline in the Participant DLQI Score at Week 12
Description: The DLQI questionnaire consists of 10 questions, where each question is scored from 0 (not affected at all) to 3 (very much affected). The DLQI score is the sum of the 10 individual question scores and ranges from 0 to 30, with lower scores indicating better quality of life. For a change from baseline, a larger negative number correlates with a greater improvement in the DLQI score.
Time Frame: Baseline and Week 12 (or end of trial if prior to Week 12)
Population: Analysis population consists of all randomized participants who received at least one dose of assigned study drug between Weeks 0 and 12 and have at least one DLQI measurement (post-baseline or baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 308 | 309 | 154
Score on a scale | -10.0 [-10.7 to -9.4] | -9.8 [-10.4 to -9.1] | -2.3 [-3.1 to -1.5]
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg (Part 1) vs Placebo (Part 1); Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; Terms for time, the interaction of time by treatment, body weight (<=90 kg, >90 kg), and prior exposure to biologic therapy for psoriasis (yes/no); Difference in least squares means = -7.7, 95% CI 2-sided [-8.6 to -6.8]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg (Part 1) vs Placebo (Part 1); Test type: Other; p < 0.001, Constrained Longitudinal Data Analysis; [statistical method as in outcome 9, analysis 1]; Difference in least squares means = -7.4, 95% CI 2-sided [-8.3 to -6.5]

10. Secondary Outcome: Percentage of Participants With DLQI Score of 0 or 1 at Week 12
Description: as for outcome 8
Time Frame: Week 12 (or end of trial if prior to Week 12)
Population: Analysis population consists of all randomized participants who received at least one dose of assigned study drug between Weeks 0 and 12 and have a DLQI measurement at Week 12 (or end of trial if prior to Week 12).
Measure: Number; unit: Percentage of participants
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1)
Number analyzed (Participants) | 299 | 304 | 150
Percentage of participants | 44.2 | 41.5 | 5.3
Statistical Analysis 1: Comparison: Tildrakizumab 200 mg (Part 1) vs Placebo (Part 1); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 38.9, 95% CI 2-sided [31.9 to 45.4]
Statistical Analysis 2: Comparison: Tildrakizumab 100 mg (Part 1) vs Placebo (Part 1); Test type: Other; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 1, analysis 1]; Difference in percentages = 36.1, 95% CI 2-sided [29.3 to 42.5]

ADVERSE EVENTS:
Time Frame: Up to 84 weeks including a 20-week follow-up period (Part 1: Week 0 to Week 12; Part 2: Week 12 to Week 28; Part 3, Week 28 to Week 64)
Description: Part 1 includes all randomized participants who received at least 1 dose of Part 1 study drug, based on the treatment received. Part 2 includes all randomized participants who received at least 1 dose of Part 2 study drug, based on the treatment received, including those on placebo re-randomized at Week 12 to tildrakizumab. Part 3 includes all participants who received at least 1 dose of Part 3 study drug, based on the treatment received, including those re-randomized to placebo during Part 3.
Groups:
- Tildrakizumab 200 mg (Part 1): Tildrakizumab 200 mg administered once a week at Weeks 0 and 4.
- Tildrakizumab 100 mg (Part 1): Tildrakizumab 100 mg administered once a week at Weeks 0 and 4.
- Placebo (Part 1): Placebo administered once a week at Weeks 0 and 4.
- Tildrakizumab 200 mg (Part 2): Tildrakizumab 200 mg administered once a week at Week 16 (includes placebo participants re-randomized at Week 12 to receive tildrakizumab 200 mg).
- Tildrakizumab 100 mg (Part 2): Tildrakizumab 100 mg administered once a week at Week 16 (includes placebo participants re-randomized at Week 12 to receive tildrakizumab 100 mg). Includes 1 participant who did not enter Part 2, but received an unscheduled dose at Week 12.
- Tildrakizumab 200 mg (Part 3): Participants received tildrakizumab 200 mg (depending on their PASI response) at Weeks 28, 40, 52, and 64 (includes participants re-randomized to placebo during Part 3).
- Tildrakizumab 100 mg (Part 3): Participants received tildrakizumab 100 mg (depending on their PASI response) at Weeks 28, 40, 52, and 64 (includes participants re-randomized to placebo during Part 3).
Arm/Group | Tildrakizumab 200 mg (Part 1) | Tildrakizumab 100 mg (Part 1) | Placebo (Part 1) | Tildrakizumab 200 mg (Part 2) | Tildrakizumab 100 mg (Part 2) | Tildrakizumab 200 mg (Part 3) | Tildrakizumab 100 mg (Part 3)
All-Cause Mortality (participants affected / at risk) | 0/308 | 0/309 | 0/155 | 0/298 | 0/299 | 0/279 | 1/19
Serious Adverse Events (participants affected / at risk) | 8/308 | 5/309 | 1/154 | 8/370 | 7/374 | 21/360 | 14/316
Other Adverse Events (participants affected / at risk) | 35/308 | 36/309 | 23/154 | 38/370 | 42/374 | 86/360 | 78/316
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tildrakizumab 200 mg (Part 1) (N=308) | Tildrakizumab 100 mg (Part 1) (N=309) | Placebo (Part 1) (N=154) | Tildrakizumab 200 mg (Part 2) (N=370) | Tildrakizumab 100 mg (Part 2) (N=374) | Tildrakizumab 200 mg (Part 3) (N=360) | Tildrakizumab 100 mg (Part 3) (N=316)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Salivary gland enlargement (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Epiglottitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Suicide attempt (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (3)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 2 (2)
Lacunar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Macular fibrosis (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis salmonella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Benign biliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Carcinoma in situ of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebellar infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Uterine haemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tildrakizumab 200 mg (Part 1) (N=308) | Tildrakizumab 100 mg (Part 1) (N=309) | Placebo (Part 1) (N=154) | Tildrakizumab 200 mg (Part 2) (N=370) | Tildrakizumab 100 mg (Part 2) (N=374) | Tildrakizumab 200 mg (Part 3) (N=360) | Tildrakizumab 100 mg (Part 3) (N=316)
Nasopharyngitis (Infections and infestations) | 20 (20) | 24 (26) | 8 (8) | 17 (18) | 24 (24) | 44 (55) | 48 (66)
Psoriasis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 8 (8) | 3 (4) | 2 (2) | 9 (9) | 9 (9)
Upper respiratory tract infection (Infections and infestations) | 15 (15) | 10 (10) | 9 (10) | 20 (21) | 16 (17) | 37 (43) | 26 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator agrees not to publish or publicly present any interim results of the trial without the prior written consent of the sponsor. The investigator further agrees to provide to the sponsor 45 days prior to submission for publication or presentation, review copies of abstracts or manuscripts for publication that report any results of the trial.